CLINICAL TRIAL: NCT03933384
Title: Tenofovir Alafenamide Versus Entecavir for the Treatment of Chronic Hepatitis B: an Open Label, Randomized Controlled Trial
Brief Title: Tenofovir Alafenamide Versus Entecavir for the Treatment of Chronic Hepatitis B
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Teng-Yu Lee, Principal Investigator, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CF18341A; 106DHA0500150 (Other Grant/Funding Number: Taichung Veterans General Hospital, Taiwan)
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis B; Viral Hepatitis
Keywords: Hepatitis B; Viral Hepatitis; Tenofovir alafenamide; Entecavir
MeSH Terms: conditions — Hepatitis B | interventions — tenofovir alafenamide; entecavir

STUDY DESIGN:
Intervention Model Description: This is a study designed for non-inferior outcome comparisons for TAF and ETV. The eligible chronic hepatitis B patients are randomly assigned (1:1) to receive once-daily oral doses of TAF 25 mg or ETV 0.5mg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tenofovir alafenamide group (Active Comparator): Study subjects will receive tenofovir alafenamide 25 mg/tab once daily
  Interventions: Drug: Tenofovir alafenamide
- Entecavir group (Active Comparator): Study subjects will receive entecavir 0.5 mg/tab once daily
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Tenofovir alafenamide — Tenofovir alafenamide 25mg/tab once daily
  Other Names: Vemlidy
  Arms: Tenofovir alafenamide group
Drug: Entecavir — Entecavir 0.5mg/tab once daily
  Other Names: Baraclude
  Arms: Entecavir group

SUMMARY:
To compare the efficacy and renal safety of tenofovir alafenamide (TAF) versus entecavir (ETV) in the chronic hepatitis B patients.

DETAILED DESCRIPTION:
With high antiviral potency and low drug resistance rate, both ETV and tenofovir disoproxil fumarate (TDF) have been recommended as the first-line antiviral therapy for chronic hepatitis B (CHB). However, risk of renal dysfunction remains an issue in TDF long-term therapy. Tenofovir alafenamide (TAF) is a novel prodrug of tenofovir and is formulated to deliver the active metabolite to target cells more efficiently than TDF at lower doses, thereby reducing systemic exposure to tenofovir. Importantly, TAF had improved renal safety as compared to TDF. TAF has been approved for treating CHB since 2017; however, it is still unknown whether the efficacy and renal safety of TAF is compatible to those of ETV. The investigators aim to conduct an open label, randomized controlled trial comparing TAF with ETV for assessing their efficacy and renal safety in CHB patients. The eligible CHB patients are randomly assigned (1:1) to receive TAF or ETV. After allocation to TAF group or ETV group, study subjects will receive therapy for 3 years (144 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Patients more than 20 years old
2. Chronic hepatitis B patients
3. Patients who were indicated for hepatitis B virus antiviral therapy

Exclusion Criteria:

1. Decompensated liver disease (Child-Pugh B &C)
2. End stage renal disease (eGRF < 15 ml/min/1.73m2)
3. Prior use of nucleot(s)ide analogues for chronic hepatitis B
4. Prior use of interferon for chronic hepatitis B within six months
5. Known history of human immunodeficiency virus or hepatitis C virus co-infection
6. Concurrent other uncontrolled malignancy
7. Women in pregnancy or lactation
8. Cannot conform to the study protocol of this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
HBV viral suppression | After 48-week therapy of Tenofovir alafenamide or entecavir
  proportion of patients with hepatitis B virus(HBV) -DNA suppression
Renal safety: Change of estimated glomerular filtration rate | After 48-week therapy of Tenofovir alafenamide or entecavir
  Change of estimated glomerular filtration rate

SECONDARY OUTCOMES:
Renal safety: Change of estimated glomerular filtration rate | After 144-week therapy of Tenofovir alafenamide or entecavir
  Change of estimated glomerular filtration rate
HBV viral suppression | After 144-week therapy of Tenofovir alafenamide or entecavir
  proportion of patients with hepatitis B virus(HBV) -DNA suppression
Normalization alanine aminotransferase (ALT) | After 144-week therapy of Tenofovir alafenamide or entecavir
  proportion of patients with ALT normalization
HBsAg loss | After 144-week therapy of Tenofovir alafenamide or entecavir
  proportion of patients with HBsAg loss
Bone mineral density | After 144-week therapy of Tenofovir alafenamide or entecavir
  change of bone mineral density

CONTACTS AND LOCATIONS:
Overall Officials: Teng-Yu Lee, MD, PhD, Study Chair — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perz JF, Armstrong GL, Farrington LA, Hutin YJ, Bell BP. The contributions of hepatitis B virus and hepatitis C virus infections to cirrhosis and primary liver cancer worldwide. J Hepatol. 2006 Oct;45(4):529-38. doi: 10.1016/j.jhep.2006.05.013. Epub 2006 Jun 23. PMID 16879891
- [Background] Chen DS, Sung JL. Hepatitis B virus infection on Taiwan. N Engl J Med. 1977 Sep 22;297(12):668-9. doi: 10.1056/NEJM197709222971213. No abstract available. PMID 757978
- [Background] Ni YH, Chang MH, Wu JF, Hsu HY, Chen HL, Chen DS. Minimization of hepatitis B infection by a 25-year universal vaccination program. J Hepatol. 2012 Oct;57(4):730-5. doi: 10.1016/j.jhep.2012.05.021. Epub 2012 Jun 2. PMID 22668640
- [Background] Chiang CJ, Yang YW, Chen JD, You SL, Yang HI, Lee MH, Lai MS, Chen CJ. Significant reduction in end-stage liver diseases burden through the national viral hepatitis therapy program in Taiwan. Hepatology. 2015 Apr;61(4):1154-62. doi: 10.1002/hep.27630. Epub 2015 Feb 10. PMID 25476749
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Kang L, Pan J, Wu J, Hu J, Sun Q, Tang J. Anti-HBV Drugs: Progress, Unmet Needs, and New Hope. Viruses. 2015 Sep 15;7(9):4960-77. doi: 10.3390/v7092854. PMID 26389937
- [Background] Lai CL, Shouval D, Lok AS, Chang TT, Cheinquer H, Goodman Z, DeHertogh D, Wilber R, Zink RC, Cross A, Colonno R, Fernandes L; BEHoLD AI463027 Study Group. Entecavir versus lamivudine for patients with HBeAg-negative chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1011-20. doi: 10.1056/NEJMoa051287. PMID 16525138
- [Background] Marcellin P, Heathcote EJ, Buti M, Gane E, de Man RA, Krastev Z, Germanidis G, Lee SS, Flisiak R, Kaita K, Manns M, Kotzev I, Tchernev K, Buggisch P, Weilert F, Kurdas OO, Shiffman ML, Trinh H, Washington MK, Sorbel J, Anderson J, Snow-Lampart A, Mondou E, Quinn J, Rousseau F. Tenofovir disoproxil fumarate versus adefovir dipivoxil for chronic hepatitis B. N Engl J Med. 2008 Dec 4;359(23):2442-55. doi: 10.1056/NEJMoa0802878. PMID 19052126
- [Background] van Bommel F, Wunsche T, Mauss S, Reinke P, Bergk A, Schurmann D, Wiedenmann B, Berg T. Comparison of adefovir and tenofovir in the treatment of lamivudine-resistant hepatitis B virus infection. Hepatology. 2004 Dec;40(6):1421-5. doi: 10.1002/hep.20464. PMID 15565615
- [Background] Tsai HJ, Chuang YW, Lee SW, Wu CY, Yeh HZ, Lee TY. Using the chronic kidney disease guidelines to evaluate the renal safety of tenofovir disoproxil fumarate in hepatitis B patients. Aliment Pharmacol Ther. 2018 Jun;47(12):1673-1681. doi: 10.1111/apt.14682. Epub 2018 Apr 25. PMID 29696665
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Chan HL, Fung S, Seto WK, Chuang WL, Chen CY, Kim HJ, Hui AJ, Janssen HL, Chowdhury A, Tsang TY, Mehta R, Gane E, Flaherty JF, Massetto B, Gaggar A, Kitrinos KM, Lin L, Subramanian GM, McHutchison JG, Lim YS, Acharya SK, Agarwal K; GS-US-320-0110 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of HBeAg-positive chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):185-195. doi: 10.1016/S2468-1253(16)30024-3. Epub 2016 Sep 22. PMID 28404091
- [Background] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092